CLINICAL TRIAL: NCT05000424
Title: Clary Sage Essential Oil Inhalation and Third Trimester Quality of Life: A Randomized, Double Blind, Controlled Trial
Brief Title: Clary Sage Essential Oil & Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nutraceuticals Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Pro00055623
Record Dates: First submitted 2021-07-26; First posted 2021-08-11 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Quality of Life; Pregnancy Related
Keywords: clary sage; essential oil; aromatherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in this group will receive a fragrant plant based massage oil with the addition of clary sage essential oil. The massage oil will be massaged into the upper thighs daily for the duration of the third trimester.
  Interventions: Other: Clary Sage Massage Oil
- Control (Placebo Comparator): Participants in this group will receive a fragrant plant based massage oil. The massage oil will be massaged into the upper thighs daily for the duration of the third trimester.
  Interventions: Other: Inert Massage Oil

INTERVENTIONS:
Other: Clary Sage Massage Oil — This massage oil contains clary sage oil. Five drops will be used daily.
  Arms: Intervention
Other: Inert Massage Oil — This massage oil consists entirely of plant based oils. Five drops will be used daily.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the potential for clary sage essential oil to support overall health, wellbeing, and quality of life during the third trimester of pregnancy among otherwise healthy adult women.

DETAILED DESCRIPTION:
Women will be informed of the opportunity to participate through their care providers, childbirth educators, or doulas. If they meet inclusion criteria, they will be given a brochure describing the risks and benefits of the study and the informed consent paperwork.

If they provide consent, they will be randomized to one of two groups: active essential oil and inert placebo. Both groups will receive a 4-ounce bottle of oil to apply daily during the third trimester of pregnancy. Those in the placebo group will be given an inert plant oil. Those in the intervention group will be given the same oil with the addition of clary sage essential oil.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-39
* Lives in the United States
* Pregnant, singleton
* Low risk
* Less than 27 weeks gestation

Exclusion Criteria:

* PCOS diagnosis
* Uncontrolled Hypertension (i.e. systolic/diastolic blood pressure > 140/90)
* Gestational Diabetes
* History of Preeclampsia
* Preterm labor
* Incompetent cervix
* Allergy to salvia sclarea or related plants
* Known Birth Defects
* Thyroid Disease diagnosis

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in salivary estriol levels from pregnancy week 27 to pregnancy week 36. | Pregnancy week 27 and 36
  salivary estriol levels are collected via the passive drool method and laboratory analyzed
Change in quality of life from week 27 to 36 of the pregnancy using the World Health Organization's Quality of Life, Brief-Form Scale (WHOQOL-BREF). | Pregnancy week 27 and 36
  This one survey measures overall quality of life through. It contains 26 questions across 4 domains. Questions are scored on a 1-5 likert scale with higher scores indicating higher quality of life.

SECONDARY OUTCOMES:
Duration of Pregnancy | from enrollment to birth, up to 16 weeks
  The total length of the pregnancy (in days) from last menstrual period to birth.
Duration of phase 2 of labor | from the onset of labor to birth, up to 24 hours
  The total length of phase 2 of labor (in minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- Franklin Health Research Center, Franklin, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No